CLINICAL TRIAL: NCT05272176
Title: Targeted Intensive Case Management of Veterans at Risk of Suicide Post Inpatient Hospitalization
Brief Title: Veterans Coordinated Community Care (3C) Study
Acronym: 3C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Harvard University (Other); Canandaigua VA Medical Center (U.S. Federal Agency); West Virginia University (Other); The Warren Alpert Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2109003096
Record Dates: First submitted 2022-01-27; First posted 2022-03-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Suicide
Keywords: Veterans; Suicide Prevention; Behavioral Symptoms; Case Management
MeSH Terms: conditions — Suicide; Suicide Prevention; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coping Long Term with Active Suicide Program (CLASP) (Experimental): The CLASP intervention is an adjunctive, telehealth-based behavioral intervention designed to reduce suicidal behavior among individuals at high risk for suicide going through periods of transition. CLASP is designed to intervene on four risk factor targets: ongoing treatment engagement, problem-solving, social and family support, and hopelessness. In addition to these general factors, the CLASP provider also has the flexibility to identify and target certain "patient-specific" risk factors (e.g., substance misuse) for intervention.
  CLASP will begin after completion of the baseline assessment, and will continue for 6 months post-discharge. CLASP will be comprised of: a) 3 initial sessions while participants are still inpatients (can occur post-discharge if needed); b) 12 brief telehealth sessions over 6-months post-discharge; c) 6 brief SO telehealth sessions.
  Interventions: Behavioral: Coping Long Term with Active Suicide Program (CLASP)
- Treatment As Usual (TAU) (No Intervention): Treatment As Usual (TAU) consists of unrestricted treatment provided as part of routine care in the Veterans Health Administration (VHA) following inpatient hospitalization. Study staff will provide no additional treatment in this arm.

INTERVENTIONS:
Behavioral: Coping Long Term with Active Suicide Program (CLASP) — Telehealth-based case management intervention designed to reduce suicidal behavior among individuals at high risk for suicide across the transition from inpatient hospitalization to the community.
  Arms: Coping Long Term with Active Suicide Program (CLASP)

SUMMARY:
Veterans Coordinated Community Care (3C) Study will recruit 850 Veterans at risk for suicide post inpatient hospitalization. Each participant will be randomly assigned to treatment as usual (TAU) or TAU plus the Coping Long Term with Active Suicide Program (CLASP), with follow-up for 6 months after discharge. Outcomes include suicide-related behaviors (including deaths due to suicide, opioid overdose, or other substance-related accidents; and nonfatal suicide attempts) and suicidal ideation and functioning.

DETAILED DESCRIPTION:
Suicide is a problem of great public health importance. The great majority of suicides occur among people with psychiatric disorders, and among psychiatric patients, those recently discharged from psychiatric hospitalization have highest suicide risk. Intensive post-discharge case management programs have been shown to reduce post-discharge suicides, but the rarity of these events even among recently-hospitalized patients makes it infeasible to argue for universal implementation of intensive post-discharge case management. Researchers propose to address this problem by carrying out a pragmatic trial among psychiatric inpatients in the Veterans Health Administration (VHA) healthcare system judged to be at high risk of post-discharge suicide (based on a validated prediction model). Researchers will evaluate the effects of a scalable remote post-discharge moderate intensity adjunctive intervention, the Coping Long Term with Active Suicide Program (CLASP), and carry out a heterogeneity of treatment effects (HTE) analysis to determine how these effects vary as a function of patient characteristics and features of the post-discharge treatment environment. Patients in the CLASP treatment will be asked to nominate a significant other (SO) to participate in the program with them. SO participation is optional. The aim of this research is to conduct a multi-site randomized controlled trial (N=850) of the CLASP intervention compared to treatment as usual for Veterans at risk for suicide post inpatient hospitalization. Assessments will occur at baseline and 6 months post discharge. Medical, administrative, and vital records will be obtained for each participant. The primary outcome of this study will be post-discharge suicide-related behaviors (including deaths due to suicide, opioid overdose, or other substance-related accidents; and nonfatal suicide attempts) in the 6 months post-discharge. Researchers will also evaluate secondary outcomes involving patient suicidal ideation and functioning.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient Veteran at high-risk for post-discharge suicide (as flagged by the study's validated prediction model)
* 18 years or older
* Access to a telephone after discharge.

Exclusion Criteria:

* Impaired decision-making capacity
* Limited or no English language proficiency
* Terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Veterans Affairs Healthcare System (VAHS) health and administrative records on suicide related behaviors | 6 months after discharge
  Suicide related behaviors that include deaths due to suicide, opioid overdose, or other substance-related accidents; and nonfatal suicide attempts.
3C Suicide Outcome Measure | 6 months after discharge
  Study specific aggregate measure (3C Suicide Outcome Measure) containing selected items from the Columbia-Suicide Severity Rating Scale (C-SSRS), Self-Injurious Thoughts and Behaviors Interview (SITBI), and Suicidal Behaviors Questionnaire (SBQ).

SECONDARY OUTCOMES:
Veterans Affairs Healthcare System (VAHS) health and administrative records on suicidal ideation and functioning | 6 months after discharge
  Suicidal ideation and functioning identified through VAHS health and administrative records
3C Suicidal Ideation and Functioning Outcome Measure | 6 months after discharge
  Study specific aggregate measure (3C Suicidal Ideation and Functioning Outcome Measure) containing selected items from the Columbia-Suicide Severity Rating Scale (C-SSRS), Self-Injurious Thoughts and Behaviors Interview (SITBI), and Suicidal Behaviors Questionnaire (SBQ), P4 Screener, Suicide Attempt Beliefs Scale (SABS), Brief Reasons for Living Inventory 10-Item Version (BRFL-10), Suicide-Related Coping Scale, and Acquired Capability for Suicide Scale

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Weinstock, PhD, Principal Investigator — Brown University
Locations (7):
- United States (7):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - VA Boston Healthcare System, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - VA St. Louis Health Care System, St Louis, Missouri
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - VA Tennessee Valley Health Care System, Murfreesboro, Tennessee
  - VA North Texas Healthcare System, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be made available through the Inter-university Consortium for Political and Social Research (ICPSR) after the study has ended.
Time Frame: De-identified data will become available after the study has ended.
Access Criteria: De-identified data are made available to users at ICPSR member institutions.

REFERENCES:
- [Background] Miller IW, Gaudiano BA, Weinstock LM. The Coping Long Term with Active Suicide Program: Description and Pilot Data. Suicide Life Threat Behav. 2016 Dec;46(6):752-761. doi: 10.1111/sltb.12247. Epub 2016 Apr 2. PMID 27038050
- [Background] Kessler RC, Bauer MS, Bishop TM, Demler OV, Dobscha SK, Gildea SM, Goulet JL, Karras E, Kreyenbuhl J, Landes SJ, Liu H, Luedtke AR, Mair P, McAuliffe WHB, Nock M, Petukhova M, Pigeon WR, Sampson NA, Smoller JW, Weinstock LM, Bossarte RM. Using Administrative Data to Predict Suicide After Psychiatric Hospitalization in the Veterans Health Administration System. Front Psychiatry. 2020 May 6;11:390. doi: 10.3389/fpsyt.2020.00390. eCollection 2020. PMID 32435212
- [Background] Miller IW, Camargo CA Jr, Arias SA, Sullivan AF, Allen MH, Goldstein AB, Manton AP, Espinola JA, Jones R, Hasegawa K, Boudreaux ED; ED-SAFE Investigators. Suicide Prevention in an Emergency Department Population: The ED-SAFE Study. JAMA Psychiatry. 2017 Jun 1;74(6):563-570. doi: 10.1001/jamapsychiatry.2017.0678. PMID 28456130
- [Derived] Weinstock LM, Bishop TM, Bauer MS, Benware J, Bossarte RM, Bradley J, Dobscha SK, Gibbs J, Gildea SM, Graves H, Haas G, House S, Kennedy CJ, Landes SJ, Liu H, Luedtke A, Marx BP, Miller A, Nock MK, Owen RR, Pigeon WR, Sampson NA, Santiago-Colon A, Shivakumar G, Urosevic S, Kessler RC. Design of a multicenter randomized controlled trial of a post-discharge suicide prevention intervention for high-risk psychiatric inpatients: The Veterans Coordinated Community Care Study. Int J Methods Psychiatr Res. 2024 Dec;33(4):e70003. doi: 10.1002/mpr.70003. PMID 39352173